CLINICAL TRIAL: NCT03107143
Title: A Randomized, Non-blind Study of TurnCare's Q-2 System on the Sacral Pressure Ulcer Prevention in High Risk Patients at St. Vincent's Medical Center
Brief Title: Study of TurnCare's Q-2 System on the Sacral Pressure Ulcer Prevention in High Risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TurnCare Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-307
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Pressure Ulcer, Buttock
Keywords: Pressure ulcer prevention; Pressure injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: A prospective, non-blinded, randomized trial. This cohort was divided into two groups: Control and Treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment Group (Experimental): Trial subjects have Q2 System installed on their beds in addition to receiving standard care of pressure ulcer prevention according to study hospital's policy and protocol.
  Interventions: Device: Q2 System
- Control Group (No Intervention): Control subjects receive only standard care of pressure ulcer prevention according to study hospital's policy and protocol without Q2 System

INTERVENTIONS:
Device: Q2 System
  Arms: Treatment Group

SUMMARY:
This is a non-blind randomized clinical trial to determine the efficacy of the TurnCare Q2 System for the prevention of sacral region (sacral, coccygeal, and buttocks) pressure ulcers. TurnCare Q2 System has 2 main components: 1. An Inflatable Skin Perfusion Enhancement Surface and 2. An Adaptive Pressure Controller. The Skin Perfusion Enhancement Surface has a patented design that accommodate human anatomy in the sacra region. The Adaptive Pressure Controller is powered by APSAR technology that provides patient specific pressure relieve in the sacral region.

DETAILED DESCRIPTION:
This study is a prospective, non-blinded randomized clinical trial. The study protocol and the consent form were approved by the IRB at the study institution. Consecutive adult patients admitted to the hospital with Braden Scale scores of 16 or less who did not meet exclusion criteria were consented and enrolled in the study. All in-patients were either scheduled admissions or were admitted through the emergency department. Upon admission, risk assessments for pressure ulcers and total body surveys were performed by the hospital staff. A Braden Scale score was determined for each patient by the hospital staff according to standard hospital protocol. Both the control group and the treatment group patients received standard care for pressure ulcer prevention according to hospital protocols, policies and guidelines. Standard pressure ulcer prevention measures for this facility include a methodology referred to as a "S.K.I.N." Bundle (S-surface selection, K-keep turning, I-incontinence management, N-nutrition.) This successful pressure ulcer prevention initiative was developed within the parent health organization and standardized throughout its 131 hospitals. In accordance with the S.K.I.N. Bundle, all patients admitted to the study hospital were repositioned every two hours, provided incontinence care, and given aggressive nutritional management as indicated. All care measures were documented in the hospital's electronic medical record (EMR) system. After obtaining informed consents, patients in the treatment group had the Q2 System placed on their beds and chairs. Perfusion enhancement surfaces were placed directly on hospital beds under the fitted bed sheets and were secured to bed frames with disposable Velcro straps. A disposable "chux" pad and lifter sheet were placed on top of the fitted sheets as is standard in most hospital settings. Adaptive pressure controllers were secured to bed footboards or attached to bases of IV poles. Specific settings for each patient were entered into the controllers. The controller settings entered included patient body weight and bed position (degrees of incline). The bed position included a bed setting (30 degrees incline) and a chair setting (90 degrees incline). When applicable, a second perfusion enhancement surface was placed on a hospital chair so that the Q2 solution could be utilized in a "sitting mode" while patients were sitting in hospital chairs. The Q2 Systems remained in continuous operation during the trial period. Patient skin did not contact any part of the Q2 system directly at any time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have a Braden Score of 16 or less without pre-existing sacral region pressure ulcers and are not subject to exclusion criteria

Exclusion Criteria:

* Pre-existing sacral region pressure ulcer
* Refusal to participate
* Inability to obtain consent
* Pregnancy
* Age less than 18 years
* Mentally challenged
* Prisoner
* Unstable spine or pelvic injuries
* Recent surgical skin graft to sacral area
* Weight > 400 lbs.
* Psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hospital acquired sacral region pressure ulcers in treatment and control groups. | Up to 10 weeks. Average of 4 weeks from enrollment.
  Rate of hospital acquired sacral pressure ulcer occurrence measurred in metrics named "number of incidences in 1,000 patient days."

CONTACTS AND LOCATIONS:
Overall Officials: Jitendra Bharucha, MD, Principal Investigator — St. Vincent's Center for Wound Healing

IPD SHARING:
Plan to Share IPD: No